CLINICAL TRIAL: NCT00953394
Title: Continuous 5-fluorouracil Infusion Plus Long Acting Octreotide in Advanced Well Differentiated Neuroendocrine Carcinomas. A Phase II Trial of the Piemonte Oncology Network.
Brief Title: 5FU and Octreotide Long-acting Release (LAR) for Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Alfredo Berruti, Dipartimento di Scienze Cliniche e Biologiche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2004-003963-58
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Neuroendocrine Tumors
Keywords: octreotide LAR; neuroendocrine carcinoma; metronomic 5fluorouracil
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment arm (Experimental): continuous 5 fluouracil infusion plus long-acting octreotide
  Interventions: Drug: continuous 5 fluouracil infusion plus long-acting octreotide

INTERVENTIONS:
Drug: continuous 5 fluouracil infusion plus long-acting octreotide — long-acting octreotide acetate at a dose of 20 mg was administered intramuscularly every 4 weeks. 5fluorouracil was given as a protracted continuous infusion without interruption at a daily dose of 200 mg/m2 of body-surface area through an elastomeric pump connected to a central venous access.
  Other Names: metronomic 5 fluouracil infusion plus long-acting octreotide

SUMMARY:
Well differentiated neuroendocrine carcinomas have low proliferative activity and conventional chemotherapy is not recommended. Metronomic chemotherapy, i.e. the frequent administration of cytotoxic drugs at low doses, has demonstrated antiangiogenetic properties. Since well differentiated NE carcinomas are highly vascular, there is a rationale for testing metronomic chemotherapy in this clinical setting.

A phase II study was designed to test the activity of protracted 5-fluorouracil (5FU) infusion plus long-acting release (LAR) octreotide for patients with neuroendocrine carcinoma.

DETAILED DESCRIPTION:
Metastatic or locally advanced well differentiated neuroendocrine carcinoma were treated with 5Fluorouracil protracted intravenous infusion (200 mg/m2 daily) plus Octreotide LAR (20 mg monthly).

Primary Endpoint: the response to treatment, evaluated according to the RECIST criteria.

Secondary Endpoints:

* toxicity, graded according to the NCI-CTG criteria;
* symptomatic response: evaluated according to the changes in both the frequency and intensity of symptoms;
* biochemical response: evaluated considering the changes in the tumor marker levels (circulating Chromogranin A);
* time to progression and survival: were measured from the date of treatment start to the date of progression and the date of last follow-up or death, respectively.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of well-differentiated neuroendocrine carcinoma according to the World Health Organization (WHO) classification;
* locally advanced or metastatic disease not amenable to surgery with radical intent;
* at least one measurable target lesion;
* radiological documentation of progressive disease;
* ECOG performance status grade <=2;
* life expectancy >12 weeks;
* adequate bone marrow reserve;
* adequate hepatic and renal function;
* ability to comply with the protocol procedures (including geographic accessibility);
* written informed consent.

Exclusion Criteria:

* non-malignant systemic disease or conditions that precluded patients from receiving the study therapy;
* second primary malignancies and previous systemic antineoplastic treatment including somatostatin analogues;
* history of prior malignancy, excepted for cured non-melanoma skin cancer, and cured in situ cervical carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-02; Primary Completion 2006-02 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
disease free survival | 50 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, PHD, Study Chair — Medical oncology, Department of Clinical and Biological Sciences, University of Turin; Luigi Dogliotti, PHD, Study Director — Medical oncology, Department of Clinical and Biological Sciences, University of Turin; Libero Ciuffreda, MD, Principal Investigator — Centro Oncologico Ematologico Subalpino, Azienda Ospedaliera Molinette, Torino
Locations (7):
- Italy (7):
  - Federico Castiglione, Alba, Cuneo
  - Davide Perroni, Saluzzo, Cuneo
  - Benedetta Ferretti, San Severino Marche, Macerata
  - Sebastiano Bombaci, Ivrea, Torino
  - Anna Ferrero, Orbassano, Torino
  - Oscar Alabiso, Novara
  - Enrica Milanesi, Torino

REFERENCES:
- [Derived] Brizzi MP, Berruti A, Ferrero A, Milanesi E, Volante M, Castiglione F, Birocco N, Bombaci S, Perroni D, Ferretti B, Alabiso O, Ciuffreda L, Bertetto O, Papotti M, Dogliotti L. Continuous 5-fluorouracil infusion plus long acting octreotide in advanced well-differentiated neuroendocrine carcinomas. A phase II trial of the Piemonte oncology network. BMC Cancer. 2009 Nov 3;9:388. doi: 10.1186/1471-2407-9-388. PMID 19886987